CLINICAL TRIAL: NCT00046813
Title: High-Dose Versus Regular-Dose Nicotine Patch for Nicotine Dependence in Individuals With Schizophrenia or Schizoaffective Disorder
Brief Title: Nicotine Patch for Nicotine Dependence in Individuals With Schizophrenia or Schizoaffective Disorder - 1
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Interim data analysis showed no effect between treatment groups
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Jill Williams, UMDNJ-Robert Wood Johnson Medical School
Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-14009-1; K23-14009-1
Record Dates: First submitted 2002-10-03; First posted 2002-10-03 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2008-08

CONDITIONS: Tobacco Use Disorder
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Tobacco Use Cessation Devices

INTERVENTIONS:
Drug: Nicotine patch

SUMMARY:
The purpose of this study is to test the use of High-Dose versus Regular-Dose Nicotine Patch for Nicotine Dependence in Individuals with Schizophrenia or Schizoaffective Disorder

DETAILED DESCRIPTION:
This is a randomized double-blind placebo controlled 8 week outpatient medication clinical trial to evaluate the relative efficacy of High-Dose (42mg) versus Regular Dose (21mg) nicotine patch treatment for individuals with schizophrenia or schizoaffective disorder and nicotine dependence. It also has a placebo controlled continuation phase to examine if longer duration of treatment is more effective than a standard eight week dosing schedule. The literature supports that schizophrenics have an increased rates of smoking and are more likely to be dependent on nicotine. Nicotine gum and patches are safe and now approved for over the counter sale in the United States. High dose patch therapy is well tolerated and provides more complete nicotine replacement. This improves withdrawal symptom relief and it is hypothesized that abstinence rates from smoking will be greater in the high dose patch group. Few trials have examined the usefulness of nicotine replacement therapy in this population and preliminary evidence shows lower than expected success rates of smoking cessation with conventional treatments

ELIGIBILITY:
Inclusion Criteria:

Subjects: 100 stable outpatients with schizophrenia and schizoaffective disorder and nicotine dependence. All subjects will meet the following inclusion criteria:

* Patients who are able to provide informed consent
* Patients will meet DSM-IV diagnostic criteria for Nicotine Dependence and Schizophrenia or Schizoaffective disorder
* Patients will be stable on their current antipsychotic regimen and will be interested in treatment for both their psychiatric and nicotine dependence

Exclusion Criteria:

* Potential subjects meeting the following criteria will be excluded:
* Patients with history of clinically significant angina or unstable angina pectoris
* Patients with severe CAD or recent myocardial infarction (within last 6 months)
* Patients with evidence or history of other severe medical illness (hematologic, renal or neoplastic)
* Patients who represent a serious suicide risk, including recent suicidal behavior or attempt within the last thirty days
* Patients with history of severe skin allergies or chronic dermatoses
* Concomitant use of clonidine or bupropion
* Pregnant females

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2001-08; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
continuous abstinence from smoking | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jill M. Williams, M.D., Principal Investigator — Rutgers, The State University of New Jersey
Locations (2):
- United States (2):
  - UMDNJ - Robert Wood Johnson Medical School-2, Piscataway, New Jersey
  - UMDNJ - Robert Wood Johnson Medical School, Piscataway, New Jersey

REFERENCES:
- [Derived] Theodoulou A, Chepkin SC, Ye W, Fanshawe TR, Bullen C, Hartmann-Boyce J, Livingstone-Banks J, Hajizadeh A, Lindson N. Different doses, durations and modes of delivery of nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2023 Jun 19;6(6):CD013308. doi: 10.1002/14651858.CD013308.pub2. PMID 37335995